CLINICAL TRIAL: NCT04147962
Title: Intense Pulsed Light in Meibomian Gland Dysfunctions: Retrospective Study
Brief Title: Intense Pulsed Light in Meibomian Gland Dysfunctions
Acronym: LACRYSTIM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Quantel Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IRBN672019/CHUSTE
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: intense pulsed light
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with dry eye disease with meibomian gland dysfunction: Collected data from patient records for consultations Day 0, Day 15 and Day 45 (3 treatment sessions) and Months 3, Months 6 (follow-up consultations).
  - parameters used for each treatment session: duration of treatment session and intensity of intense pulsed light
  Interventions: Device: intense pulsed light (usual practice)

INTERVENTIONS:
Device: intense pulsed light (usual practice) — collection data : parameters used for each treatment session: duration of treatment session and intensity of intense pulsed light

SUMMARY:
Dry eye disease (DED) is an extremely common disease whose meibomian gland dysfunction is the main etiology.

Polychromatic intense pulsed light (IPL) is a promising new therapeutic alternative but few clinical data have been published.

A new IPL device has recently been marketed: LACRYSTIM (QUANTEL, France). The investigators have been using it in our clinical practice since June 2019.

The investigators present a retrospective study on our first clinical results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Dry eye disease with meibomian gland dysfunction, preferentially mild to moderate, and having benefited from intense pulsed light treatment.
* patient affiliated with a social security organization

Exclusion Criteria:

* patient with incomplete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Dry eye disease with meibomian gland dysfunction, preferentially mild to moderate, and having benefited from intense pulsed light treatment
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Lacrydiag in current clinical practice | 6 months
  The LacryDiag ocular surface analyzer is used for the diagnosis of dry eyes.

SECONDARY OUTCOMES:
collection of adverse events | 6 months
  -data concerning the safety: presence or absence of adverse events during treatment or afterwards (burns, tingling, redness of skin ...)
Ocular Surface Disease Index questionnaire | 6 months
  measured in current clinical practice. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers.
Slit lamp Photography x16 and x25 | 6 months
  in current clinical practice
Oxford Score | 6 months
  measured in current clinical practice. The Oxford score is used to assess epithelial damage to the cornea and conjunctiva.
Break-up time Test | 6 months
  measured in current clinical practice. The measurement of the tear film rupture time determines the stability of the tear film, i.e. the degree of humidification of the eyes.
Schirmer Test | 6 months
  measured in current clinical practice. Determination of the quantity of tears produced.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caroline TRONE, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trone MC, Garcin T, Ollier E, Thuret G, Gain P. A retrospective study of the efficacy of intense pulsed light delivered by the Lacrystim(R) for meibomian gland dysfunction therapy. BMC Ophthalmol. 2022 Aug 6;22(1):335. doi: 10.1186/s12886-022-02531-7. PMID 35933379